CLINICAL TRIAL: NCT01129479
Title: Galantamine Treatment for Nonfluent Aphasia in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Responsible Party: Heidi Roth, University of North Carolina
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GAL-EMR-4008
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia; treatment; cholinesterase inhibitor; stroke
MeSH Terms: conditions — Aphasia; Stroke | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Galantamine (Active Comparator)
  Interventions: Drug: Galantamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Galantamine — Galantamine XL 8 mg for 4 weeks, followed by Galantamine XL 16 mg for subsequent 12 weeks. Taken in the morning with food for total of 12 weeks.
  Other Names: Razadyne; Reminyl
  Arms: Galantamine
Drug: Placebo pill — Placebo pill each morning with food for 12 weeks.
  Arms: Placebo

SUMMARY:
Cognitive impairment after stroke is common and has a major effect on morbidity and quality of life. Acetylcholinesterase inhibitors have demonstrated benefit in vascular dementia, but efficacy in treating more circumscribed cognitive deficits following stroke, such as aphasia, has not been systematically investigated.

This study evaluated the efficacy of Galantamine (Reminyl) in subjects with chronic, stable non-fluent aphasia secondary to stroke. Subjects enrolled in a double-blind placebo- controlled cross-over study that employed a comprehensive battery of language tests and measures of general cognitive and behavioral status that will be used to control for factors that may influence language functioning. The primary study outcome was a within-subject comparison of changes in language function and behavioral scores between placebo and active-treatment phases (12 weeks each). Our hypothesis was that by increasing acetylcholine levels, and facilitating activity of other neurotransmitters affecting attentional systems, Galantamine would produce gains in both language and behavioral scores in patients suffering chronic effects in cognitive systems due to injury following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of aphasia with relatively spared comprehension.
* Onset 6 months or greater prior to enrollment.
* Native English speaker
* Right-handed.
* Adults (18 years of age or older).

Exclusion Criteria:

* Patients receiving ongoing individual speech therapy. (Most patients are no longer eligible for individualized speech therapy after 6 months from stroke onset, thus this should not eliminate many patients).
* Extremely mild or extremely severe aphasia. (Boston Naming Test Score <3 or >45 items named from 60 items).
* Global dementia (and any other patient with reduced decisional capacity requiring a legally authorized representative for consent).
* Presence of major cognitive deficit other than aphasia caused by stroke related disease.
* Contraindications to cholinomimetic agents: History of active peptic ulcer disease within 1 year, Severe asthma, unstable angina, bradyarrhythmia with resting pulse less than 50, sick sinus syndrome, or seizures.
* Major psychiatric disorders that affect cognition including: psychosis, major depression, bipolar disorder, alcohol or substance abuse.
* Major medical conditions that alter cognition (e.g., heart failure, dialysis dependent renal failure, hepatic failure, active cancer).
* Impairments that affect metabolism of the medication including: Severe renal impairment (Creatinine clearance equal to or greater than 9), and moderate or severe hepatic impairment (Child-Pugh score >7)
* Patients using medications that have major effects on brain neurotransmitter systems or cognition within 2 months of enrollment. Exclusionary medications are: medications with significant anti-cholinergic activity (tricyclic antidepressants, diphenhydramine), anti-Parkinsonian medications (including Sinemet, amantadine, bromocriptine, pergolide, selegiline), and narcotic analgesics (> 2 doses per week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Spontaneous Speech | Every 4 weeks
  Analysis of spontaneous speech production with picture description (cookie theft picture): content units and lexical efficiency; as well as Boston Naming Test naming latency.

SECONDARY OUTCOMES:
ADP | Every 4 weeks
  Aphasia Diagnostic Profile: lexical Retrieval, phrase length, phonemic fluency, and category fluency.
Communication Log scores | Every 12 weeks
  Subject communication change log scores Caregiver communication change log score

CONTACTS AND LOCATIONS:
Overall Officials: Heidi L Roth, MD, Principal Investigator — University of North Carolina